CLINICAL TRIAL: NCT06796777
Title: Residual Paralysis in the Post Anesthesia Care Unit: the Association Beetween Residual Neuromuscular Block Risk Prediction Score and the Train-of-Four Ratio. a Prospective Single-Center Open-Label Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Mostafa kamel Mohamed, residant doctor, Assiut University
Other Study IDs: NMB RPS Train four ratio
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Residual Paralysis
Keywords: Residual Neuromuscular Block Risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients who will be scheduled to undergo elective surgical procedures requiring the use of neuromus

SUMMARY:
The reported incidence of rNMB varies between 16% to more than 70 depending on the used definition (train-of-four [TOF] ratio 0.7 or 0.9), type of NMBA, type of reversal agent, and timing of measurements The degree of residual paralysis can be evaluated in different ways: clinical tests requiring the patients cooperation, which normally can be performed only after emergence; visual or tactile evaluation of responses to TOF or double-burst stimulation (DBS) at the adductor pollicis (qualitative or subjective assessment); and measurement of the TOF ratio (TOFr) with a device (quantitative or objective measurement), For several years, the standard criterion for adequate neuromuscular function recovery was a TOF ratio of 0.7 Residual paralysis risk prediction score (REPS) has been recently invented to identify surgical patients who might be at an increased risk for the development of rNMB. Ten independent predictors for residual paralysis were identified and used for the score development.

Recent literature reported that REPS ≥4 is significantly associated with an increased risk of postoperative respiratory complications when neuromuscular monitoring is not used Does of reverse is neostigmine(.04-.08)mg/kg and does of Atropine .01mg /kg Time of surgical intervention not affecte measurement of residual paralysis in PACU the aim of the study evaluate the degree of association, and the predictive accuracy of the REPS (as a predictive tool) compared with the TOFr as a quantitative assessment tool for (rNMB) in surgical patients in the early postoperative phase. The TOFr will be measured at 0, 15, 30, 45, and 60 min after extubation.

DETAILED DESCRIPTION:
The reported incidence of rNMB varies between 16% to more than 70 depending on the used definition (train-of-four [TOF] ratio 0.7 or 0.9), type of NMBA, type of reversal agent, and timing of measurements The degree of residual paralysis can be evaluated in different ways: clinical tests requiring the patients cooperation, which normally can be performed only after emergence; visual or tactile evaluation of responses to TOF or double-burst stimulation (DBS) at the adductor pollicis (qualitative or subjective assessment); and measurement of the TOF ratio (TOFr) with a device (quantitative or objective measurement), For several years, the standard criterion for adequate neuromuscular function recovery was a TOF ratio of 0.7 Residual paralysis risk prediction score (REPS) has been recently invented to identify surgical patients who might be at an increased risk for the development of rNMB. Ten independent predictors for residual paralysis were identified and used for the score development.

Recent literature reported that REPS ≥4 is significantly associated with an increased risk of postoperative respiratory complications when neuromuscular monitoring is not used Does of reverse is neostigmine(.04-.08)mg/kg and does of Atropine .01mg /kg Time of surgical intervention not affecte measurement of residual paralysis in PACU the aim of the study evaluate the degree of association, and the predictive accuracy of the REPS (as a predictive tool) compared with the TOFr as a quantitative assessment tool for (rNMB) in surgical patients in the early postoperative phase. The TOFr will be measured at 0, 15, 30, 45, and 60 min after extubation.

ELIGIBILITY:
Inclusion Criteria:

- 1- Age group 18-65 years old 2- Both genders 3- Patients who will be scheduled to undergo elective surgical procedures requiring the use of neuromuscular blocking drugs.

5- Patients with American Society of Anesthesiologist physical status classification of 1 or 2.

Exclusion Criteria:

* 1- Patients who are less than 18 years old or more than 65 years old. 2- Patients with planned scheduled recovery in the intensive care unit or if more than 10 minutes had elapsed since tracheal extubation until NMB monitoring at the PACU.

  3- Patients on medications that interfere with muscle activity. 4- Known allergy to neuromuscular blocking agents. 5- Pregnancy or suspected pregnancy. 6- Neuro-muscular diseases. 7- Patients refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be scheduled to undergo elective surgical procedures requiring the use of neuromuscular blocking drugs.
Sampling Method: Probability Sample
Enrollment: 91 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of residual neuromascular block | 60 minutes
  the incidence of rNMB assessed by train-of-four ratio at admission to the PACU and at 15, 30, 45, and 60 min after PACU admission to be correlated with the Risk Prediction Score

IPD SHARING:
Plan to Share IPD: Undecided